CLINICAL TRIAL: NCT06169514
Title: Understanding the Health Systems and Policy Contexts of Medical Oxygen in Africa and Asia (MOXY-HSP)
Brief Title: Health Systems and Policy Contexts of Medical Oxygen
Acronym: MOXY-HSP
Status: Recruiting | Type: Observational
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: University of Ibadan (Other); University of Health Sciences, Lao People's Democratic Republic (PDR) (Unknown); University of Health Sciences, Cambodia (Unknown); Makerere University (Other); Ministry of Health, Liberia (Other); Ministry of Health, Rwanda (Other Government); Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: HREC 100143
Record Dates: First submitted 2023-10-29; First posted 2023-12-13 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-11

CONDITIONS: Hypoxemia; Morality; Pneumonia
Keywords: Health system; Oxygen; Oxygen systems; Oxygen access; Pulse oximetry
MeSH Terms: conditions — Hypoxia; Pneumonia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Policy and stakeholder analysis across 6 countries: Policy and stakeholder analysis across 6 countries
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This is a mixed-methods program evaluation from a health systems and policy perspective, involving (i) stakeholder analysis, (ii) policy-implementation gap analysis, and (iii) comparative country case studies. This study aims to understand how national oxygen strategies achieve impact at national, and subnational level, across country contexts, at what cost.

The the investigators seek to:

1. Involve policymakers, implementers (including private sector), and medical oxygen users in identifying challenges and understanding potential solutions to medical oxygen access;
2. Generate new data on how medical oxygen systems work and can be improved from multiple perspectives;
3. Draw lessons on medical oxygen that can directly inform national and global practice and policy.

This study will be conducted in 6 of the 9 countries participating in the Clinton Health Access Initiative (CHAI) led Medical Oxygen Implementation (MOXY) program (Uganda, Nigeria, Rwanda, Liberia, Lao PDR, Cambodia).

Key informants will be selected representing government, non-governmental agencies, professional associations, private sector, and civil society. This study will be completed over 4 years, with timelines varying between country study sites.

DETAILED DESCRIPTION:
The investigators will use a concurrent mixed-methods design, with an overarching comparative case study methodology. The investigators will adopt an iterative approach, using co-design to adapt the study methodology to the specific context of each country and annual learning team meetings with stakeholders to refine the final case study topics (sub-study 3) and methodology.

Three embedded sub-studies are planned:

Sub-study 1 (Stakeholder Analysis) aims to understand the policy environment for medical oxygen services across different country contexts. This will be informed by the MOXY baseline survey, which includes data on oxygen-related facility readiness and clinical practices across the MOXY program areas. Data sources will include stakeholder interviews with participants from different levels (national, provincial, local) and policy perspectives (government, implementing/advising partners, practitioners, beneficiaries). Results will inform sub-study 2 and MOXY program implementation.

Sub-study 2 (Policy-Implementation Gap Analysis) aims to critically analyse the gap between policy intentions and actual implementation. This will be informed by the baseline facility readiness and clinical practice data. Data sources will include a desk review of oxygen-related policies, stakeholder in-depth interviews, and program administrative data. Results will inform implementation of country oxygen strategies and feed into prioritization of focus areas for sub-study 3.

Sub-study 3 (Comparative Country Case Studies) aims to compare oxygen programs across countries, focusing on particular challenges or unique solutions identified in sub-study 1 and 2. Data sources will include repeated desk review of oxygen-related policies and program administrative data, follow-up stakeholder interviews, and triangulation with quantitative survey results on facility readiness and clinical practices.

This research will also draw on national stakeholder dialogues - both to review, refine, and validate preliminary findings of the study team and to draw out feasible solutions/alternatives for both policy and practice and oxygen eco-system. In year 1 the investigators will generate key evidence about how the current strategies and polices are being translated into action, identifying key opportunities for implementing partners to focus support. Over years 2 and 3, the investigators will learn how these activities have affected medical oxygen service coverage, drawing lessons across country contexts and across different implementation approaches.

ELIGIBILITY:
Key informants will be selected representing government, non-governmental agencies, professional associations, private sector, and civil society.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted in 6 of the 9 countries participating in the CHAI-led MOXY program (Uganda, Nigeria, Rwanda, Liberia, Lao PDR, Cambodia).
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
In-depth stakeholder interviews on national medical oxygen strategies | 4 years
  In depth stakeholder interviews covering perspectives on policies, oversight, implementation, and related support towards the particular domain (e.g. measurement and indicators, health workforce capacity building, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Hamish Graham, PhD, Principal Investigator — Murdoch Childrens Research Institute; Carina King, PhD, Principal Investigator — Karolinska Institutet
Locations (6):
- Cambodia, Phnom Penh, Cambodia
- Lao PDR, Vientiane, Laos
- Liberia, Monrovia, Liberia
- Nigeria, Ibadan, Nigeria
- Rwanda, Kigali, Rwanda
- Uganda, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No